CLINICAL TRIAL: NCT01517984
Title: Immune Monitoring and Calcineurin Inhibitor (CNI) Withdrawal in Low Risk Recipients of Kidney Transplantation
Brief Title: Immune Monitoring and CNI Withdrawal in Low Risk Recipients of Kidney Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Absence of equipoise on the basis of predetermined stopping rules.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Clinical Trials in Organ Transplantation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CTOT-09
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Results first posted 2016-11-30 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-08

CONDITIONS: Kidney Transplant Recipients
Keywords: recipients of living-donor kidney allografts; antithymocyte globulin (ATG) induction; calcineurin inhibitors (CNIs); CNI withdrawal
MeSH Terms: interventions — Tacrolimus; cni protein, Drosophila; Prednisone; thymoglobulin; Calcineurin Inhibitors; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus (CNI) Withdrawal (Experimental): Subjects randomized (2:1) to tacrolimus (CNI) withdrawal.
  Recipients of living-donor kidney allografts are given induction therapy with rabbit antithymocyte globulin (RATG, Thymoglobulin®) and treated with a standard immunosuppressive regimen of mycophenolate mofetil (MMF), prednisone and tacrolimus.Subjects without any clinical acute rejection (AR) in the first 6 months, without borderline or acute rejection on the 6 month biopsy, and without donor-specific antibody (DSA) at anytime, including the 6 month test are randomized (2:1) to tacrolimus (CNI) withdrawal.
  Interventions: Drug: Tacrolimus (CNI) Withdrawal; Drug: Standard Immunosuppressive Therapy
- Standard Immunosuppressive Therapy (Active Comparator): Subjects randomized to standard immunosuppressive therapy, without subsequent tacrolimus (CNI) withdrawal.
  Recipients of living-donor kidney allografts are given induction therapy with rabbit antithymocyte globulin (RATG, Thymoglobulin®) and treated with a standard immunosuppressive regimen of mycophenolate mofetil (MMF), prednisone and tacrolimus. Tacrolimus (CNI) withdrawal does not occur.
  Interventions: Drug: Standard Immunosuppressive Therapy

INTERVENTIONS:
Drug: Tacrolimus (CNI) Withdrawal — Recipients of living-donor kidney allografts are given induction therapy with rabbit antithymocyte globulin (RATG, Thymoglobulin®) and treated with a regimen of mycophenolate mofetil (MMF), prednisone and tacrolimus.
  Subjects without any clinical acute rejection (AR) in the first 6 months, without borderline or acute rejection on the 6 month biopsy, and without donor-specific antibody (DSA) at anytime, including the 6 month test will be randomized (2:1) to tacrolimus (CNI) withdrawal.
  Other Names: ATG Induction,Tacrolimus (CNI), MMF and Prednisone, Followed by CNI Withdrawal; rabbit antithymocyte globulin (RATG); Thymoglobulin®; calcineurin inhibitor (CNI); mycophenolate mofetil; CellCept®
  Arms: Tacrolimus (CNI) Withdrawal
Drug: Standard Immunosuppressive Therapy — Recipients of living-donor kidney allografts are given induction therapy with rabbit antithymocyte globulin (RATG, Thymoglobulin®) and treated with a regimen of mycophenolate mofetil (MMF), prednisone and tacrolimus.
  Other Names: ATG induction,Tacrolimus (CNI), MMF and Prednisone; rabbit antithymocyte globulin (RATG); Thymoglobulin®; calcineurin inhibitor (CNI); mycophenolate mofetil; CellCept®

SUMMARY:
The study will compare how well transplanted kidneys work and the response of people's immune systems as tacrolimus, a calcineurin inhibitor (CNI), is withdrawn. In addition, this research study will evaluate whether reducing immunosuppression can decrease some of these side effects while still preventing rejection of the kidney.

DETAILED DESCRIPTION:
Kidney transplantation is a treatment option for people with kidney disease. However, there is still much to learn about how to best care for the transplanted kidney and keep it functioning for a long time. Transplant recipients take immunosuppression (anti-rejection) drugs to prevent their body from rejecting the new kidney. These drugs are used to prevent the immune system from attacking the transplanted kidney. All anti-rejection medications have unwanted side effects. The purpose of this study is to evaluate the safety of slowly removing tacrolimus, a CNI.

ELIGIBILITY:
INCLUSION CRITERIA -

Initial Enrollment/Screening: Patients who meet all of the following criteria are eligible for enrollment as study subjects:

* Subject must be able to understand and provide written informed consent;
* Primary living-donor (related or unrelated) kidney transplant recipients;
* Peak flow-based PRAs for class I and class II <30%(performed by local center);
* Current (within 8 weeks prior to transplantation) flow-based PRAs for class I and class II <30% (performed by local center);
* No donor specific antibody by flow solid phase method on the peak PRA serum (if serum available), or on the current PRA serum (within 8 weeks prior to transplantation) performed by central core laboratory. If the sera for the peak PRA is not available, then only the current PRA serum will be tested;
* Negative T-cell and B-cell crossmatch by flow cytometry (performed by local center);
* Female subjects of childbearing potential must have a negative pregnancy test (urine or serum) upon study entry;
* Female and male subjects with reproductive potential must agree to use FDA approved methods of birth control while participating in the study.

Inclusion Criteria for Randomization:

Participants who meet all of the following criteria are eligible for randomization:

* No history of acute rejection episodes;
* The pre-randomization protocol biopsy should confirm no rejection, including borderline rejection (based on the central pathology read);
* No donor specific antibody as detected by flow solid phase method (performed by the central core laboratory).

EXCLUSION CRITERIA -

Initial Enrollment/Screening:

Participants who meet any of these criteria are not eligible for enrollment as study subjects:

* Recipient of multiple organ transplants;
* Prior history of organ transplantation;
* Deceased-donor source;
* Any condition that would preclude protocol biopsies;
* HLA identical recipients;
* Currently breast-feeding or plans to become pregnant during the timeframe of the study follow up period;
* Any condition that, in the opinion of the investigator, would interfere with the subject's ability to comply with study requirements;
* Inability or unwillingness to comply with study protocol;
* Use of investigational drugs within 4 weeks of study entry and for the duration of the study;
* Recent recipient of any licensed or investigational live attenuated vaccine(s) within two months of prior to study entry.

Exclusion Criteria for Randomization:

Participants who meet any of these criteria are not eligible for randomization:

* Subjects who receive less than 4.5mg/kg of Rabbit ATG (Thymoglobulin®) induction therapy;
* Subjects who test positive for BKV by PCR in the blood at 6 months post-transplant;
* Any condition that would preclude protocol biopsies;
* Currently breast-feeding or plans to become pregnant during the timeframe of the study follow up period;
* Any condition that, in the opinion of the investigator, would interfere with the subject's ability to comply with study requirements;
* Inability or unwillingness of a subject to give written informed consent or comply with study protocol;
* Use of investigational drugs within 4 weeks of study entry and for the duration of the study;
* Subjects who receive less than 1500 mg daily of Mycophenolate Mofetil (CellCept®) or equivalent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Hricik, MD, Study Chair — University Hospitals Cleveland Medical Center; Peter S. Heeger, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (11):
- United States (9):
  - University of California Los Angeles, Los Angeles, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Mount Sinai School of Medicine, New York, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Methodist Hospital, Houston, Texas
- Canada (2):
  - Health Sciences Centre, Winnipeg, Manitoba
  - Toronto General Hospital, Toronto, Ontario

REFERENCES:
- [Result] Hricik DE, Formica RN, Nickerson P, Rush D, Fairchild RL, Poggio ED, Gibson IW, Wiebe C, Tinckam K, Bunnapradist S, Samaniego-Picota M, Brennan DC, Schroppel B, Gaber O, Armstrong B, Ikle D, Diop H, Bridges ND, Heeger PS; Clinical Trials in Organ Transplantation-09 Consortium. Adverse Outcomes of Tacrolimus Withdrawal in Immune-Quiescent Kidney Transplant Recipients. J Am Soc Nephrol. 2015 Dec;26(12):3114-22. doi: 10.1681/ASN.2014121234. Epub 2015 Apr 29. PMID 25925687
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Clinical Trials in Organ Transplantation (CTOT) — https://www.ctotstudies.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Enrolled, Not Transplanted: These participants were consented and enrolled into the study, but did receive a living-donor kidney allograft transplant as specified by the protocol.
- Transplanted, Not Randomized: These participants were enrolled into the study and received a living-donor kidney allograft transplant. Participants were given an induction therapy with rabbit antithymocyte globulin (1.5-2.0 mg/kg daily for 5 days) and treated with a regimen of mycophenolate mofetil (target dose of 1000 mg twice daily), prednisone (no less than 5 mg/day or 10 mg every other day) and tacrolimus (0.1 mg/kg twice daily, adjusted to target trough levels of 8-12 ng/ml in first 3 months post-transplant, 5-8 ng/ml thereafter). Participants were followed for up to 8 months and deemed ineligible for randomization or terminated for other reasons.
- Randomized to Tacrolimus Withdrawal: These participants were enrolled into the study and received a living-donor kidney allograft transplant. Participants were given an induction therapy with rabbit antithymocyte globulin (1.5-2.0 mg/kg daily for 5 days) and treated with a regimen of mycophenolate mofetil (target dose of 1000 mg twice daily), prednisone (no less than 5 mg/day or 10 mg every other day) and tacrolimus (0.1 mg/kg twice daily, adjusted to target trough levels of 8-12 ng/ml in first 3 months post-transplant, 5-8 ng/ml thereafter). Participants were followed for 6-8 months then randomized to tacrolimus withdrawal. Following randomization these participants had their dose of tacrolimus withdrawn gradually over three to four months, with complete withdrawal occurring no later than four months. Participants were followed up to 18 months after being randomized.
- Randomized to Control Group: Participants were given an induction therapy with rabbit antithymocyte globulin (1.5-2.0 mg/kg daily for 5 days) and treated with a regimen of mycophenolate mofetil (target dose of 1000 mg twice daily), prednisone (no less than 5 mg/day or 10 mg every other day) and tacrolimus (0.1 mg/kg twice daily, adjusted to target trough levels of 8-12 ng/ml in first 3 months post-transplant, 5-8 ng/ml thereafter). Participants were followed for 6-8 months then randomized to control group, where they continued on the pre-randomization standard care of mycophenolate mofetil, prednisone, and tacrolimus. Participants were followed up to 18 months after being randomized.
Period: Overall Study
Arm/Group | Enrolled, Not Transplanted | Transplanted, Not Randomized | Randomized to Tacrolimus Withdrawal | Randomized to Control Group
Started | 5 | 26 | 14 | 7
Completed | 0 | 3 | 10 | 6
Not Completed | 5 | 23 | 4 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 8 | 4 | 1
Not completed — Screen Failure | 4 | 0 | 0 | 0
Not completed — Ineligible for randomization | 0 | 14 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Transplanted, But Not Randomized: These participants were enrolled into the study and received a living-donor kidney allograft transplant. Participants were given an induction therapy with rabbit antithymocyte globulin (1.5-2.0 mg/kg daily for 5 days) and treated with a regimen of mycophenolate mofetil (target dose of 1000 mg twice daily), prednisone (no less than 5 mg/day or 10 mg every other day) and tacrolimus (0.1 mg/kg twice daily, adjusted to target trough levels of 8-12 ng/ml in first 3 months post-transplant, 5-8 ng/ml thereafter). Participants were followed for up to 8 months and deemed ineligible for randomization or terminated for other reasons.
- Randomized to Control Group: Participants were given an induction therapy with rabbit antithymocyte globulin (1.5-2.0 mg/kg daily for 5 days) and treated with a regimen of mycophenolate mofetil (target dose of 1000 mg twice daily), prednisone (no less than 5 mg/day or 10 mg every other day) and tacrolimus (0.1 mg/kg twice daily, adjusted to target trough levels of 8-12 ng/ml in first 3 months post-transplant, 5-8 ng/ml thereafter). Participants were followed for 6-8 months then randomized to control group, where the continued on the pre-randomization standard care of mycophenolate mofetil, prednisone, and tacrolimus. Participants were followed up to 18 months after being randomized.
- Total: Total of all reporting groups
Arm/Group | Transplanted, But Not Randomized | Randomized to Tacrolimus Withdrawal | Randomized to Control Group | Total
Number analyzed (Participants) | 26 | 14 | 7 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (11.6) | 46.5 (14.4) | 44.9 (8.5) | 50.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 0 | 12
  Male | 20 | 8 | 7 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 0 | 4
  White | 22 | 10 | 7 | 39
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 4 | 0 | 7
  United States | 23 | 10 | 7 | 40
HLA mismatch [Mean (Standard Deviation); unit: Number of HLA marker mismatches] — Human leukocyte antigen (HLA) is a protein - or marker - found on most cells in your body and is used to match you with a donor for your bone marrow or cord blood transplant. The best transplant outcome happens when a patient's HLA and donor's HLA closely match. There are at least 8 HLA markers that are typically compared prior to transplantation. A mismatch of greater than three indicates that there is a potential for a poorer outcome than a better HLA match between donor and recipient.
  Number of HLA marker mismatches | 3.6 (1.7) | 3.4 (1.3) | 3.4 (1.3) | 3.4 (1.4)
CMV status (donor, recipient) [Number; unit: participants] — Cytomegalovirus (CMV) is a common virus, and is a concern when a person has a weakened immune system, such as during transplantation. Once infected with CMV, your body retains the virus for life. CMV can spread from donor to recipient during transplant and dormant CMV in the recipient could become active following transplantation due to weakened immune system. CMV positive recipients have a higher likelihood for incidence of CMV disease and allograft loss.
  participants
    Donor +, Recipient + | 8 | 5 | 0 | 13
    Donor +, Recipient - | 5 | 2 | 1 | 8
    Donor -, Recipient + | 3 | 2 | 2 | 7
    Donor -, Recipient - | 9 | 5 | 3 | 17
    Donor not done, Recipient + | 0 | 0 | 1 | 1
    Donor missing, Recipient - | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Incremental IF/A Scores >2 at 24 Months Post-Randomization
Description: The investigators were not able to assess this outcome, the effect of the intervention on interstitial fibrosis/tubular atrophy (IF/TA; on a 2-year graft biopsy) due to the study's premature termination by the Data Safety Monitoring Board (DSMB) because of absence of equipoise on the basis of predetermined stopping rules.
Time Frame: IF/TA scores on protocol biopsies obtained at 24 months post-randomization will be compared to those obtained at the time of implantation for this measurement.
Population: No analyses were performed due to early study closure.
Arm/Group | Randomized to Tacrolimus Withdrawal | Randomized to Control Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Estimated GFR Using the Chronic Kidney Disease Epidemiology (CKD-EPI) Equation
Description: Estimated glomerular filtration rate (eGFR) is a test to measure the level of kidney function. In this measure, the effects of tacrolimus withdrawal on long-term kidney function was assessed by comparing absolute 24 month eGFR (18 months post-randomization) and change in eGFR from 6 to 24 months (randomization to 18 months randomization). Lower numbers indicate poorer kidney function
Time Frame: 6 months post-transplantation, 24 months post-transplantation
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Randomized to Tacrolimus Withdrawal | Randomized to Control Group
Number analyzed (Participants) | 14 | 7
mL/min
  6 Month eGFR | 56.2 (13.9) | 62.3 (15.0)
  24 Month eGFR | 61.7 (14.8) | 68.6 (24.1)
  Change in eGFR from 6 to 24 months | 5.5 (12.0) | 6.3 (12.6)

3. Secondary Outcome: Incidence of Acute Rejection
Description: Acute renal allograft rejection is defined as histological reading of borderline or greater determined by the local pathology laboratory. Participants suspected of having a rejection episode on the basis of clinical signs, symptoms, or on the basis of laboratory tests, had a renal ultrasound and underwent a renal transplant biopsy. Any detection of acute cellular rejection or acute humoral rejection resulted in participants in the 'Randomized to Tacrolimus Withdrawal' group to be restarted on tacrolimus and followed per the reduced follow-up schedule of events.
Time Frame: 6 to 18 months post-randomization
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Randomized to Tacrolimus Withdrawal | Randomized to Control Group
Number analyzed (Participants) | 14 | 7
participants | 6 | 0

4. Secondary Outcome: Allograft Survival Rate
Description: Allograft survival is defined as participants who did not need to be re-transplanted or placed on dialysis due to the failure of their allograft transplantation during the course of this study.
Time Frame: 6 to 18 months post-randomization
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Randomized to Tacrolimus Withdrawal | Randomized to Control Group
Number analyzed (Participants) | 14 | 7
participants | 14 | 7

5. Secondary Outcome: Participant Survival Rate
Description: Number of participants who did not die within the course of this study.
Time Frame: 6 to 18 months post-transplantation
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | Randomized to Tacrolimus Withdrawal | Randomized to Control Group
Number analyzed (Participants) | 14 | 7
participants | 14 | 7

6. Secondary Outcome: Percentage of Participants With New Donor Specific Antibodies (DSAs)
Description: Donor specific antibodies are antibodies that are directed against antigens expressed on donor organs. These antibodies can result in an immune attack on the transplanted organ, increasing risk of graft loss and/or rejection.
Time Frame: 6 to 18 months post-randomization
Population: Intent-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | Randomized to Tacrolimus Withdrawal | Randomized to Control Group
Number analyzed (Participants) | 14 | 7
percentage of participants | 36 | 14

7. Secondary Outcome: Percentage of Participants With Donor-Specific Memory Using Elispot
Description: This endpoint was unable to be analyzed because the study was terminated early after stopping rules were met.
Time Frame: 6 to 18 months post-randomization
Population: No analyses were performed due to early study closure.
Arm/Group | Randomized to Tacrolimus Withdrawal | Randomized to Control Group
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percentage of Participants in the Experimental Arm Off Tacrolimus
Description: Participants in the 'Randomized to Tacrolimus Withdrawal' group were considered fully withdrawn once they no longer received any doses of tacrolimus. Participants met this endpoint if they did not resume taking tacrolimus as of 18 months post randomization with stable allograft function and without rejection of donor-specific antibodies.
Time Frame: 18 months post-randomization
Population: Intent-to-treat
Measure: Number; unit: percentage of participants
Arm/Group | Randomized to Tacrolimus Withdrawal
Number analyzed (Participants) | 14
percentage of participants | 43

9. Secondary Outcome: Incremental Change in IF/TA Scores
Description: This endpoint was unable to be analyzed because the study was terminated early after stopping rules were met.
Time Frame: 6 to 18 months post-transplant
Population: No analyses were performed due to early study closure.
Arm/Group | Randomized to Tacrolimus Withdrawal | Randomized to Control Group
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Measurement of Urinary Parameters Before and After Randomization
Description: This endpoint was unable to be analyzed because the study was terminated early after stopping rules were met.
Time Frame: 6 months post-transplantation to 18 months post-randomization
Population: No analyses were performed due to early study closure.
Arm/Group | Randomized to Tacrolimus Withdrawal | Randomized to Control Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Transplantation through end of study (up to 24 months)
Arm/Group | Transplanted, But Not Randomized | Randomized to Tacrolimus Withdrawal | Randomized to Control Group
Serious Adverse Events (participants affected / at risk) | 2/26 | 4/14 | 0/7
Other Adverse Events (participants affected / at risk) | 4/26 | 5/14 | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplanted, But Not Randomized (N=26) | Randomized to Tacrolimus Withdrawal (N=14) | Randomized to Control Group (N=7)
Transplant rejection (Immune system disorders) | 1 (1) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplanted, But Not Randomized (N=26) | Randomized to Tacrolimus Withdrawal (N=14) | Randomized to Control Group (N=7)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hernia obstructive (General disorders) | 1 (1) | 0 (0) | 0 (0)
Transplant rejection (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
BK virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
After meeting protocol stopping rules, this trial was closed to new enrollment and randomization. No additional prespecified withdrawal of tacrolimus was allowed. Those already enrolled or randomized were followed for up to 24 months post-transplant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No